CLINICAL TRIAL: NCT02031354
Title: Prospective "Pre-post" Pilot Study on the Effects of Dietary Chloride Supplementation on Neurohormonal and Diuretic Function in Patients With Heart Failure
Brief Title: A Pilot Study of Dietary Chloride Supplementation on Cardiorenal Function in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1308012508
Record Dates: First submitted 2013-12-12; First posted 2014-01-09 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Heart Failure
Keywords: Lysine Chloride
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lysine Chloride (Experimental)
  Interventions: Dietary Supplement: Lysine Chloride

INTERVENTIONS:
Dietary Supplement: Lysine Chloride — Administration of 21g of lysine chloride (7g three times daily) for a period of time of 3 days

SUMMARY:
The purpose of this study is to determine if administration of supplemental chloride in the form of lysine chloride to patients with congestive heart failure will affect their neurohormonal profile as well as response to diuretics.

DETAILED DESCRIPTION:
This prospective pilot "pre-post" study was designed to determine if supplementation of sodium free chloride ion as a lysine chloride to patients with heart failure could improve parameters of neurohormonal status and diuretic responsiveness. Volunteers will receive Lysine Chloride 7 grams three times daily for three days. At baseline and then again post lysine chloride patients will undergo sampling of venous blood for determination of neurohormonal parameters in addition to formal diuretic responsiveness testing.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Fluency in English
* Heart failure requiring loop diuretic therapy
* Loop diuretic dose ≥ 80mg/day furosemide equivalents
* Stable volume status and diuretic requirement as assessed by treating physician

Exclusion Criteria:

* Unstable heart failure
* renal replacement therapy or an estimated GFR < 30 ml/min/1.73m2
* Significant bladder dysfunction
* History of hepatic failure
* Pregnancy
* History of hyperinsulinemia/hyperlysinuria

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in plasma renin activity following lysine chloride administration | 3 days
Change in urinary renin level following lysine chloride administration | 3 days
Change in diuretic response following lysine chloride administration | 3 days
  Diuretic response will me evaluated by measuring volume of urine produced following diuretic administration

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Testani, MD/MTR, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Background] Licata G, Di Pasquale P, Parrinello G, Cardinale A, Scandurra A, Follone G, Argano C, Tuttolomondo A, Paterna S. Effects of high-dose furosemide and small-volume hypertonic saline solution infusion in comparison with a high dose of furosemide as bolus in refractory congestive heart failure: long-term effects. Am Heart J. 2003 Mar;145(3):459-66. doi: 10.1067/mhj.2003.166. PMID 12660669
- [Background] Kirchner KA, Kotchen TA, Galla JH, Luke RG. Importance of chloride for acute inhibition of renin by sodium chloride. Am J Physiol. 1978 Nov;235(5):F444-50. doi: 10.1152/ajprenal.1978.235.5.F444. PMID 31796
- [Background] RUBIN AL, SPRITZ N, MEAD AW, HERRMANN RA, BRAVEMAN WS, LUCKEY EH. The use of L-lysine monomydrochloride in combination with mercurial diuretics in the treatment of refractory fluid retention. Circulation. 1960 Mar;21:332-6. doi: 10.1161/01.cir.21.3.332. No abstract available. PMID 14439868
- [Derived] Hanberg JS, Rao V, Ter Maaten JM, Laur O, Brisco MA, Perry Wilson F, Grodin JL, Assefa M, Samuel Broughton J, Planavsky NJ, Ahmad T, Bellumkonda L, Tang WH, Parikh CR, Testani JM. Hypochloremia and Diuretic Resistance in Heart Failure: Mechanistic Insights. Circ Heart Fail. 2016 Aug;9(8):10.1161/CIRCHEARTFAILURE.116.003180 e003180. doi: 10.1161/CIRCHEARTFAILURE.116.003180. PMID 27507113